CLINICAL TRIAL: NCT02247076
Title: Does Meal Timing Affect Energy Expenditure
Acronym: GRAZING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Principal Investigator, Courtney Peterson, Instructor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 2014-038
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Meal Timing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazing (Placebo Comparator): Participants will eat meals spread over the course of the day ("grazing").
  Interventions: Behavioral: Grazing
- Time-restricted feeding (early eating) (Experimental): Participants will eat meals only in the early part of the day (early lunch and very early dinner).
  Interventions: Behavioral: Time-restricted feeding (early eating)

INTERVENTIONS:
Behavioral: Grazing
  Arms: Grazing
Behavioral: Time-restricted feeding (early eating)
  Arms: Time-restricted feeding (early eating)

SUMMARY:
The purpose of this study is to find out if meal timing affects calories burned and blood sugar levels.

DETAILED DESCRIPTION:
10 overweight adult men and women will eat according to two different eating schedules: grazing and time-restricting feeding ("early eating"). While on each eating schedule, metabolism (calories burned) will be measured during a 24-hour stay in a respiratory chamber. Glucose levels-as well as key diurnal rhythms such in heart rate-will also be measured continuously. This study requires two 1-week periods of participation.

ELIGIBILITY:
Inclusion Criteria:

* Are 20-45 years of age
* Have a weight between 150 and 220 lbs
* Have a body mass index between 25 and 35 kg/m2 inclusive (a number calculated from your height and weight)
* If you are a female, have a regular menstrual cycle that is between 25 and 35 days long
* If you are female, had your period within the last 35 days
* Regularly go to sleep between 9:30 pm and 12:00 am
* Regularly eat dinner 9 or more hours after eating breakfast
* Are willing to have about 2/3 cup of your blood stored for future research related to this study

Exclusion Criteria:

* Have diabetes or are on anti-diabetes medication
* Suffer from significant cardiovascular, renal (kidney), cardiac (heart), liver, lung or nervous system disease
* Have stomach or intestinal problems
* Regularly use medications such as steroids, beta blockers, adrenergic-stimulating agents, and laxatives
* Take any medications or supplements known to affect sleep, circadian rhythms, or metabolism (with the exception that certain forms of birth control are allowed)
* Have abnormal lab work that is clinically significant in the opinion of the study physician
* Are pregnant or lactating
* Take the Depo Provera shot, or use an Interuterine Device (IUD) or hormone patch for birth control
* If you are on hormonal birth control, have been on a stable dose for less than 3 months
* Have smoked or used nicotine/tobacco products within the last 3 months
* Regularly do competitive sport training
* Perform overnight shift work an average of one or more times per week
* Have an irregular sleep schedule
* Have an irregular eating schedule
* Regularly drink 3 or more drinks of alcohol per day
* Are not able or are unwilling to eat only the food and drink served to you by Pennington Biomedical, while in the study
* Are not able or are unwilling to refrain from strenuous exercise while participating in the study
* Are not able to spend 2 separate full days (for about 25 hours each) at Pennington Biomedical
* Are not able to maintain a consistent sleep schedule while participating in the study
* Are not able to maintain a consistent eating schedule while participating in the study
* Are not able to stop drinking coffee and other caffeine-containing drinks on the day of and day prior to testing

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Energy expenditure (calories burned) | 2 days

SECONDARY OUTCOMES:
Blood sugar levels | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Peterson, PhD, MSc, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Ravussin E, Beyl RA, Poggiogalle E, Hsia DS, Peterson CM. Early Time-Restricted Feeding Reduces Appetite and Increases Fat Oxidation But Does Not Affect Energy Expenditure in Humans. Obesity (Silver Spring). 2019 Aug;27(8):1244-1254. doi: 10.1002/oby.22518. PMID 31339000